CLINICAL TRIAL: NCT02081001
Title: Comparison of Pharmacokinetic and Pharmacodynamic Profiles of G-Pump™ (Glucagon Infusion) vs. GlucaGen® Delivered Subcutaneously to Subjects With Type 1 Diabetes (T1DM)
Brief Title: PK/PD Study With G-Pump (Glucagon Infusion) in T1DM Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xeris Pharmaceuticals (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Emissary International LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: XSGO-201; 4R44DK096706-02 (NIH)
Record Dates: First submitted 2014-03-04; First posted 2014-03-07 (Estimated); Results first posted 2016-08-01 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-03

CONDITIONS: Hypoglycemia
Keywords: Hypoglycemia; Glucagon; Artificial Pancreas
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- G-Pump™ (glucagon infusion) (Experimental): G-Pump™ (glucagon infusion); single subcutaneous infusion doses at 0.3 μg/kg, 1.2 μg/kg and 2.0 μg/kg
  Interventions: Drug: Novo Nordisk GlucaGen®; Drug: G-Pump™ (glucagon infusion)
- Novo Nordisk GlucaGen® (Active Comparator): Novo Nordisk GlucaGen®; single subcutaneous infusion doses 0.3 μg/kg, 1.2 μg/kg and 2.0 μg/kg
  Interventions: Drug: Novo Nordisk GlucaGen®; Drug: G-Pump™ (glucagon infusion)

INTERVENTIONS:
Drug: Novo Nordisk GlucaGen® — single subcutaneous infusion doses at 0.3 μg/kg, 1.2 μg/kg and 2.0 μg/kg
Drug: G-Pump™ (glucagon infusion) — single subcutaneous infusion doses at 0.3 μg/kg, 1.2 μg/kg and 2.0 μg/kg

SUMMARY:
The purpose of the study is to assess the safety, speed of absorption, and onset of action of G-Pump™ (glucagon infusion) at three subcutaneous doses as compared to Novo GlucaGen®, all delivered via an OmniPod® infusion pump to patients with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Males or females diagnosed with type 1 diabetes mellitus for at least 24 months
* Current usage of subcutaneous insulin pump treatment
* Age 18-65 years
* C-peptide level < 0.5 ng/ml
* Willingness to follow all study procedures, including attending all clinic visits
* Subject has provided informed consent and has signed and dated an informed consent form before any trial-related activities

Exclusion Criteria:

* Pregnant and/ or Lactating: For women of childbearing potential: there is a requirement for a negative urine pregnancy test and for agreement to use contraception during the study and for at least 1 month after participating in the study.
* HbA1c >10.0%
* Renal insufficiency (serum creatinine of 1.2 mg/dL or greater)
* Serum ALT or AST equal to or greater than 3 times the upper limit of normal; hepatic synthetic insufficiency as defined as a serum albumin of less than 3.0 g/dL; or serum bilirubin of over 2.0.
* Hematocrit of less than or equal to 34%
* Congestive heart failure, NYHA class II, III or IV
* History of coronary artery disease
* Active foot ulceration
* History of a cerebrovascular accident
* Active alcohol abuse or substance abuse
* Active malignancy, except basal cell or squamous cell skin cancers
* Major surgical operation within 30 days prior to screening
* Seizure disorder
* Current administration of oral or parenteral corticosteroids
* Use of an investigational drug within 30 days prior to screening
* Bleeding disorder, treatment with warfarin, or platelet count below 50,000
* Proliferative or severe non-proliferative retinopathy
* Gastroparesis
* Personal or family history of pheochromocytoma or disorder with increased risk of pheochromocytoma (MEN 2, neurofibromatosis, or Von Hippel-Lindau disease)
* Insulinoma
* Allergies to glucagon or glucagon-like products, or any history of significant hypersensitivity to glucagon or any related products.
* Glycogen storage disease
* Any concurrent illness, other than diabetes, that is not controlled by a stable therapeutic regimen
* Whole blood donation of 1 pint (500 mL) within 8 weeks prior to Screening.
* Any reason the principal investigator deems exclusionary

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-03; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Castle, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 19 adults ages 18-65 years with type 1 diabetes were recruited over a period of 4 months to receive treatment at a public university hospital.
Pre-assignment Details: A total of 30 subjects were screened for study inclusion. The 19 subjects who met all eligibility criteria were randomized and assigned to treatment.
Groups:
- Dose Order: 0.3, 1.2 & 2 μg/kg; Drug Order: G-Pump/GlucaGen: Subjects received three doses of glucagon 2.5 hours apart at each of two treatment visits separated by a wash-out period of 3-28 days. Bolus doses were administered subcutaneously via an OmniPod infusion pump placed on the anterior abdomen. Subjects in this group received doses in the order of 0.3, 1.2 and 2.0 μg/kg of body weight at each visit, and received G-Pump glucagon at the first treatment visit and GlucaGen at the second treatment visit.
- Dose Order: 0.3, 1.2 & 2 μg/kg; Drug Order: GlucaGen/G-Pump: Subjects received three doses of glucagon 2.5 hours apart at each of two treatment visits separated by a wash-out period of 3-28 days. Bolus doses were administered subcutaneously via an OmniPod infusion pump placed on the anterior abdomen. Subjects in this group received doses in the order of 0.3, 1.2 and 2.0 μg/kg of body weight at each visit, and received GlucaGen at the first treatment visit and G-Pump glucagon at the second treatment visit.
- Dose Order: 0.3, 2 & 1.2 μg/kg; Drug Order: G-Pump/GlucaGen: Subjects received three doses of glucagon 2.5 hours apart at each of two treatment visits separated by a wash-out period of 3-28 days. Bolus doses were administered subcutaneously via an OmniPod infusion pump placed on the anterior abdomen. Subjects in this group received doses in the order of 0.3, 2.0 and 1.2 μg/kg of body weight at each visit, and received G-Pump glucagon at the first treatment visit and GlucaGen at the second treatment visit.
- Dose Order: 0.3, 2 & 1.2 μg/kg; Drug Order: GlucaGen/G-Pump: Subjects received three doses of glucagon 2.5 hours apart at each of two treatment visits separated by a wash-out period of 3-28 days. Bolus doses were administered subcutaneously via an OmniPod infusion pump placed on the anterior abdomen. Subjects in this group received doses in the order of 0.3, 2.0 and 1.2 μg/kg of body weight at each visit, and received GlucaGen at the first treatment visit and G-Pump glucagon at the second treatment visit.
- Dose Order: 1.2, 0.3 & 2 μg/kg; Drug Order: G-Pump/GlucaGen: Subjects received three doses of glucagon 2.5 hours apart at each of two treatment visits separated by a wash-out period of 3-28 days. Bolus doses were administered subcutaneously via an OmniPod infusion pump placed on the anterior abdomen. Subjects in this group received doses in the order of 1.2, 0.3 and 2.0 μg/kg of body weight at each visit, and received G-Pump glucagon at the first treatment visit and GlucaGen at the second treatment visit.
- Dose Order: 1.2, 0.3 & 2 μg/kg; Drug Order: GlucaGen/G-Pump: Subjects received three doses of glucagon 2.5 hours apart at each of two treatment visits separated by a wash-out period of 3-28 days. Bolus doses were administered subcutaneously via an OmniPod infusion pump placed on the anterior abdomen. Subjects in this group received doses in the order of 1.2, 0.3 and 2.0 μg/kg of body weight at each visit, and received GlucaGen at the first treatment visit and G-Pump glucagon at the second treatment visit.
- Dose Order: 1.2, 2 & 0.3 μg/kg; Drug Order: G-Pump/GlucaGen: Subjects received three doses of glucagon 2.5 hours apart at each of two treatment visits separated by a wash-out period of 3-28 days. Bolus doses were administered subcutaneously via an OmniPod infusion pump placed on the anterior abdomen. Subjects in this group received doses in the order of 1.2, 2 and 0.3 μg/kg of body weight at each visit, and received G-Pump glucagon at the first treatment visit and GlucaGen at the second treatment visit.
- Dose Order: 1.2, 2 & 0.3 μg/kg; Drug Order: GlucaGen/G-Pump: Subjects received three doses of glucagon 2.5 hours apart at each of two treatment visits separated by a wash-out period of 3-28 days. Bolus doses were administered subcutaneously via an OmniPod infusion pump placed on the anterior abdomen. Subjects in this group received doses in the order of 1.2, 2 and 0.3 μg/kg of body weight at each visit, and received GlucaGen at the first treatment visit and G-Pump glucagon at the second treatment visit.
- Dose Order: 2, 0.3 & 1.2 μg/kg; Drug Order: G-Pump/GlucaGen: Subjects received three doses of glucagon 2.5 hours apart at each of two treatment visits separated by a wash-out period of 3-28 days. Bolus doses were administered subcutaneously via an OmniPod infusion pump placed on the anterior abdomen. Subjects in this group received doses in the order of 2.0, 0.3 and 1.2 μg/kg of body weight at each visit, and received G-Pump glucagon at the first treatment visit and GlucaGen at the second treatment visit.
- Dose Order: 2, 0.3 & 1.2 μg/kg; Drug Order: GlucaGen/G-Pump: Subjects received three doses of glucagon 2.5 hours apart at each of two treatment visits separated by a wash-out period of 3-28 days. Bolus doses were administered subcutaneously via an OmniPod infusion pump placed on the anterior abdomen. Subjects in this group received doses in the order of 2.0, 0.3 and 1.2 μg/kg of body weight at each visit, and received GlucaGen at the first treatment visit and G-Pump glucagon at the second treatment visit.
- Dose Order: 2, 1.2 & 0.3 μg/kg; Drug Order: G-Pump/GlucaGen: Subjects received three doses of glucagon 2.5 hours apart at each of two treatment visits separated by a wash-out period of 3-28 days. Bolus doses were administered subcutaneously via an OmniPod infusion pump placed on the anterior abdomen. Subjects in this group received doses in the order of 2.0, 1.2 and 0.3 μg/kg of body weight at each visit, and received G-Pump glucagon at the first treatment visit and GlucaGen at the second treatment visit.
- Dose Order: 2, 1.2 & 0.3 μg/kg; Drug Order: GlucaGen/G-Pump: Subjects received three doses of glucagon 2.5 hours apart at each of two treatment visits separated by a wash-out period of 3-28 days. Bolus doses were administered subcutaneously via an OmniPod infusion pump placed on the anterior abdomen. Subjects in this group received doses in the order of 2.0, 1.2 and 0.3 μg/kg of body weight at each visit, and received GlucaGen at the first treatment visit and G-Pump glucagon at the second treatment visit.
Period: Overall Study
Arm/Group | Dose Order: 0.3, 1.2 & 2 μg/kg; Drug Order: G-Pump/GlucaGen | Dose Order: 0.3, 1.2 & 2 μg/kg; Drug Order: GlucaGen/G-Pump | Dose Order: 0.3, 2 & 1.2 μg/kg; Drug Order: G-Pump/GlucaGen | Dose Order: 0.3, 2 & 1.2 μg/kg; Drug Order: GlucaGen/G-Pump | Dose Order: 1.2, 0.3 & 2 μg/kg; Drug Order: G-Pump/GlucaGen | Dose Order: 1.2, 0.3 & 2 μg/kg; Drug Order: GlucaGen/G-Pump | Dose Order: 1.2, 2 & 0.3 μg/kg; Drug Order: G-Pump/GlucaGen | Dose Order: 1.2, 2 & 0.3 μg/kg; Drug Order: GlucaGen/G-Pump | Dose Order: 2, 0.3 & 1.2 μg/kg; Drug Order: G-Pump/GlucaGen | Dose Order: 2, 0.3 & 1.2 μg/kg; Drug Order: GlucaGen/G-Pump | Dose Order: 2, 1.2 & 0.3 μg/kg; Drug Order: G-Pump/GlucaGen | Dose Order: 2, 1.2 & 0.3 μg/kg; Drug Order: GlucaGen/G-Pump
Started | 2 | 1 | 2 | 1 | 3 | 1 | 2 | 1 | 2 | 1 | 2 | 1
Completed | 2 | 1 | 2 | 1 | 2 | 1 | 2 | 1 | 2 | 1 | 2 | 1
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized subjects
Groups:
- Xeris G-Pump Glucagon First, Followed by GlucaGen: Subjects who received G-Pump (glucagon infusion) at the first treatment visit and GlucaGen at the second treatment visit.
- GlucaGen First, Followed by Xeris G-Pump: Subjects who received GlucaGen at the first treatment visit and G-Pump (glucagon infusion) at the second treatment visit.
- Total: Total of all reporting groups
Arm/Group | Xeris G-Pump Glucagon First, Followed by GlucaGen | GlucaGen First, Followed by Xeris G-Pump | Total
Number analyzed (Participants) | 13 | 6 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 6 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (9.54) | 32.2 (8.38) | 35.3 (9.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 5 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 11 | 5 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 6 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: Time to Reach 50% of Maximum Glucose Concentration (Glucose T50%-Early)
Description: The onset of action was assessed by determining the time in minutes required to achieve 50% of the maximum plasma concentration of glucose following each dose of glucagon.
Time Frame: 0 to 150 minutes post-dosing
Population: All randomized, evaluable subjects. Two subjects not evaluable for response to GlucaGen due to dosing errors were excluded from the analysis. In addition, subjects with no increase in glucose concentration post-dosing (i.e., maximum concentration was at time zero) were not evaluable for response and consequently were not included in the analysis.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- 0.3 μg/kg G-Pump: 0.3 μg/kg dose of G-Pump (glucagon infusion) delivered via OmniPod sc infusion pump
- 1.2 μg/kg G-Pump: 1.2 μg/kg dose of G-Pump (glucagon infusion) delivered via OmniPod sc infusion pump
- 2.0 μg/kg G-Pump: 2.0 μg/kg dose of G-Pump (glucagon infusion) delivered via OmniPod sc infusion pump
- 0.3μg/kg GlucaGen: 0.3 μg/kg dose of GlucaGen delivered via OmniPod sc infusion pump
- 1.2 μg/kg GlucaGen: 1.2 μg/kg dose of GlucaGen delivered via OmniPod sc infusion pump
- 2.0 μg/kg GlucaGen: 2.0 μg/kg dose of GlucaGen delivered via OmniPod sc infusion pump
Arm/Group | 0.3 μg/kg G-Pump | 1.2 μg/kg G-Pump | 2.0 μg/kg G-Pump | 0.3μg/kg GlucaGen | 1.2 μg/kg GlucaGen | 2.0 μg/kg GlucaGen
Number analyzed (Participants) | 14 | 18 | 19 | 11 | 16 | 16
minutes | 17.2 (8.76) | 21.9 (18.44) | 21.3 (16.52) | 7.6 (9.45) | 14.5 (15.36) | 22.8 (6.51)
Statistical Analysis 1: Comparison: 0.3 μg/kg G-Pump vs 0.3μg/kg GlucaGen; Test type: Superiority or Other; p = 0.23, Mixed Models Analysis; Point estimate ratio = 2.06, 90% CI 2-sided [0.74 to 5.75], Standard Error of Mean 1.19
Statistical Analysis 2: Comparison: 1.2 μg/kg G-Pump vs 1.2 μg/kg GlucaGen; Test type: Superiority or Other; p = 0.52, Mixed Models Analysis; Point estimate ratio = 1.25, 90% CI 2-sided [0.69 to 2.28], Standard Error of Mean 0.43
Statistical Analysis 3: Comparison: 2.0 μg/kg G-Pump vs 2.0 μg/kg GlucaGen; Test type: Superiority or Other; p = 0.49, Mixed Models Analysis; Point estimate ratio = 0.86, 90% CI 2-sided [0.59 to 1.25], Standard Error of Mean 0.19

2. Primary Outcome: Time to Reach 50% of Maximum Glucagon Concentration (Glucagon T50%-Early)
Description: The speed of absorption was assessed by determining the time in minutes required to achieve 50% of the maximum plasma concentration of glucagon following each dose of glucagon.
Time Frame: 0 to 150 minutes post-dosing
Population: All randomized, evaluable subjects. Two subjects not evaluable for response to GlucaGen due to dosing errors were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- 0.3 μg/kg GlucaGen: 0.3 μg/kg dose of GlucaGen delivered via OmniPod sc infusion pump
Arm/Group | 0.3 μg/kg G-Pump | 1.2 μg/kg G-Pump | 2.0 μg/kg G-Pump | 0.3 μg/kg GlucaGen | 1.2 μg/kg GlucaGen | 2.0 μg/kg GlucaGen
Number analyzed (Participants) | 19 | 19 | 19 | 16 | 16 | 16
minutes | 12.2 (10.51) | 12.4 (5.07) | 13.9 (4.65) | 7.6 (3.51) | 10.5 (4.46) | 11.0 (3.09)
Statistical Analysis 1: Comparison: 0.3 μg/kg G-Pump vs 0.3 μg/kg GlucaGen; Test type: Superiority or Other; p = 0.23, Mixed Models Analysis; Point estimate ratio = 1.37, 90% CI 2-sided [0.88 to 2.12], Standard Error of Mean 0.34
Statistical Analysis 2: Comparison: 1.2 μg/kg G-Pump vs 1.2 μg/kg GlucaGen; Test type: Superiority or Other; p = 0.09, Mixed Models Analysis; Point estimate ratio = 1.29, 90% CI 2-sided [1.01 to 1.65], Standard Error of Mean 0.18
Statistical Analysis 3: Comparison: 2.0 μg/kg G-Pump vs 2.0 μg/kg GlucaGen; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis; Point estimate ratio = 1.36, 90% CI 2-sided [1.11 to 1.67], Standard Error of Mean 0.16

3. Secondary Outcome: Glucagon Cmax
Description: Maximum plasma concentration of glucagon
Time Frame: From 0 to 150 minutes post-dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/dl
Arm/Group | 0.3 μg/kg G-Pump | 1.2 μg/kg G-Pump | 2.0 μg/kg G-Pump | 0.3 μg/kg GlucaGen | 1.2 μg/kg GlucaGen | 2.0 μg/kg GlucaGen
Number analyzed (Participants) | 19 | 19 | 19 | 16 | 16 | 16
pg/dl | 168.1 (57.66) | 328.2 (127.9) | 440.6 (310.9) | 140.2 (53.69) | 229.3 (161.6) | 446.9 (220.4)
Statistical Analysis 1: Comparison: 0.3 μg/kg G-Pump vs 0.3 μg/kg GlucaGen; Test type: Superiority or Other; p = 0.15, Mixed Models Analysis; Point estimate ratio = 1.26, 90% CI 2-sided [0.97 to 1.64], Standard Error of Mean 0.19
Statistical Analysis 2: Comparison: 1.2 μg/kg G-Pump vs 1.2 μg/kg GlucaGen; Test type: Superiority or Other; p = 0.24, Mixed Models Analysis; Point estimate ratio = 1.29, 90% CI 2-sided [0.90 to 1.84], Standard Error of Mean 0.26
Statistical Analysis 3: Comparison: 2.0 μg/kg G-Pump vs 2.0 μg/kg GlucaGen; Test type: Superiority or Other; p = 0.31, Mixed Models Analysis; Point estimate ratio = 0.83, 90% CI 2-sided [0.60 to 1.14], Standard Error of Mean 0.15

4. Secondary Outcome: Glucose Cmax
Description: Maximum plasma concentration of glucose
Time Frame: From 0 to 150 minutes post-dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | 0.3 μg/kg G-Pump | 1.2 μg/kg G-Pump | 2.0 μg/kg G-Pump | 0.3 μg/kg GlucaGen | 1.2 μg/kg GlucaGen | 2.0 μg/kg GlucaGen
Number analyzed (Participants) | 19 | 19 | 19 | 16 | 16 | 16
mg/dl | 177.6 (43.1) | 198.8 (49.37) | 212.6 (57.18) | 162.0 (51.69) | 183.3 (66.15) | 200.6 (63.81)
Statistical Analysis 1: Comparison: 0.3 μg/kg G-Pump vs 0.3 μg/kg GlucaGen; Test type: Superiority or Other; p = 0.09, Mixed Models Analysis; Point estimate ratio = 1.18, 90% CI 2-sided [1.01 to 1.39], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: 1.2 μg/kg G-Pump vs 1.2 μg/kg GlucaGen; Test type: Superiority or Other; p = 0.29, Mixed Models Analysis; Point estimate ratio = 1.12, 90% CI 2-sided [0.93 to 1.35], Standard Error of Mean 0.12
Statistical Analysis 3: Comparison: 2.0 μg/kg G-Pump vs 2.0 μg/kg GlucaGen; Test type: Superiority or Other; p = 0.24, Mixed Models Analysis; Point estimate ratio = 1.11, 90% CI 2-sided [0.96 to 1.28], Standard Error of Mean 0.09

5. Secondary Outcome: Glucagon Tmax
Description: Time to maximum plasma concentration of glucagon
Time Frame: From 0 to 150 minutes post-dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 0.3 μg/kg G-Pump | 1.2 μg/kg G-Pump | 2.0 μg/kg G-Pump | 0.3 μg/kg GlucaGen | 1.2 μg/kg GlucaGen | 2.0 μg/kg GlucaGen
Number analyzed (Participants) | 19 | 19 | 19 | 16 | 16 | 16
minutes | 24.5 (23.42) | 27.3 (12.93) | 31.9 (15.93) | 23.3 (10.71) | 23.9 (6.31) | 23.9 (8.74)
Statistical Analysis 1: Comparison: 0.3 μg/kg G-Pump vs 0.3 μg/kg GlucaGen; Test type: Superiority or Other; p = 0.70, Mixed Models Analysis; Point estimate ratio = 0.91, 90% CI 2-sided [0.60 to 1.38], Standard Error of Mean 0.22
Statistical Analysis 2: Comparison: 1.2 μg/kg G-Pump vs 1.2 μg/kg GlucaGen; Test type: Superiority or Other; p = 0.19, Mixed Models Analysis; Point estimate ratio = 1.26, 90% CI 2-sided [0.94 to 1.68], Standard Error of Mean 0.21
Statistical Analysis 3: Comparison: 2.0 μg/kg G-Pump vs 2.0 μg/kg GlucaGen; Test type: Superiority or Other; p = 0.052, Mixed Models Analysis; Point estmate ratio = 1.45, 90% CI 2-sided [1.07 to 1.98], Standard Error of Mean 0.26

6. Secondary Outcome: Glucose Tmax
Description: Time to maximum plasma concentration of glucose
Time Frame: From 0 to 150 minutes post-dosing
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 0.3 μg/kg G-Pump | 1.2 μg/kg G-Pump | 2.0 μg/kg G-Pump | 0.3 μg/kg GlucaGen | 1.2 μg/kg GlucaGen | 2.0 μg/kg GlucaGen
Number analyzed (Participants) | 14 | 18 | 19 | 11 | 16 | 16
minutes | 38.2 (29.62) | 49.5 (41.79) | 49.4 (40.59) | 25.9 (28.38) | 31.2 (34.75) | 52.8 (20.21)
Statistical Analysis 1: Comparison: 0.3 μg/kg G-Pump vs 0.3 μg/kg GlucaGen; Test type: Superiority or Other; p = 0.16, Mixed Models Analysis; Point estimate ratio = 2.02, 90% CI 2-sided [0.87 to 4.66], Standard Error of Mean 0.95
Statistical Analysis 2: Comparison: 1.2 μg/kg G-Pump vs 1.2 μg/kg GlucaGen; Test type: Superiority or Other; p = 0.48, Mixed Models Analysis; Point estimate ratio = 1.31, 90% CI 2-sided [0.68 to 2.54], Standard Error of Mean 0.49
Statistical Analysis 3: Comparison: 2.0 μg/kg G-Pump vs 2.0 μg/kg GlucaGen; Test type: Superiority or Other; p = 0.28, Mixed Models Analysis; Point estimate ratio = 0.80, 90% CI 2-sided [0.57 to 1.13], Standard Error of Mean 0.16

7. Secondary Outcome: Glucagon AUC
Description: Area under the plasma concentration time curve for glucagon
Time Frame: From 0 to 150 minutes post-dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: (pg/dl)*minutes
Arm/Group | 0.3 μg/kg G-Pump | 1.2 μg/kg G-Pump | 2.0 μg/kg G-Pump | 0.3 μg/kg GlucaGen | 1.2 μg/kg GlucaGen | 2.0 μg/kg GlucaGen
Number analyzed (Participants) | 19 | 19 | 19 | 16 | 16 | 16
(pg/dl)*minutes | 12104 (3944) | 21177 (6139) | 27595 (14530) | 11070 (3032) | 15781 (7874) | 27355 (10757)
Statistical Analysis 1: Comparison: 0.3 μg/kg G-Pump vs 0.3 μg/kg GlucaGen; Test type: Superiority or Other; p = 0.61, Mixed Models Analysis; Point estimate ratio = 1.06, 90% CI 2-sided [0.87 to 1.30], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: 1.2 μg/kg G-Pump vs 1.2 μg/kg GlucaGen; Test type: Superiority or Other; p = 0.22, Mixed Models Analysis; Point estimate ratio = 1.19, 90% CI 2-sided [0.94 to 1.5], Standard Error of Mean 0.16
Statistical Analysis 3: Comparison: 2.0 μg/kg G-Pump vs 2.0 μg/kg GlucaGen; Test type: Superiority or Other; p = 0.26, Mixed Models Analysis; Point estimate ratio = 0.84, 90% CI 2-sided [0.66 to 1.09], Standard Error of Mean 0.12

8. Secondary Outcome: Glucose AUC
Description: Area under the plasma concentration time curve for glucose
Time Frame: From 0 to 150 minutes post-dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: (mg/dl)*minutes
Arm/Group | 0.3 μg/kg G-Pump | 1.2 μg/kg G-Pump | 2.0 μg/kg G-Pump | 0.3 μg/kg GlucaGen | 1.2 μg/kg GlucaGen | 2.0 μg/kg GlucaGen
Number analyzed (Participants) | 19 | 19 | 19 | 16 | 16 | 16
(mg/dl)*minutes | 22296 (7998) | 26251 (7110) | 27360 (8190) | 21005 (7931) | 24079 (9348) | 25845 (8624)
Statistical Analysis 1: Comparison: 0.3 μg/kg G-Pump vs 0.3 μg/kg GlucaGen; Test type: Superiority or Other; p = 0.19, Mixed Models Analysis; Point estimate ratio = 1.18, 90% CI 2-sided [0.96 to 1.46], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: 1.2 μg/kg G-Pump vs 1.2 μg/kg GlucaGen; Test type: Superiority or Other; p = 0.21, Regression, Cox; Point estimate ratio = 1.15, 90% CI 2-sided [0.95 to 1.38], Standard Error of Mean 0.12
Statistical Analysis 3: Comparison: 2.0 μg/kg G-Pump vs 2.0 μg/kg GlucaGen; Test type: Superiority or Other; p = 0.19, Mixed Models Analysis; Point estimate ratio = 1.13, 90% CI 2-sided [0.97 to 1.31], Standard Error of Mean 0.10

9. Secondary Outcome: Infusion Site Discomfort Score at 10 Minutes
Description: Infusion site discomfort was assessed by the subjects using a 100 mm Visual Analog Scale (VAS) questionnaire at 10 minutes following the initiation of dosing. Subjects were asked to draw a vertical line across the horizontal scale to indicate their current level of discomfort from 0 = no discomfort to 100 = worst possible discomfort. The distance in mm from the left hand anchor to the the first point where the subject's mark crossed the horizontal scale was measured and reported as the infusion site discomfort score.
Time Frame: At 10 minutes post-dosing
Population: All treated subjects
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0.3 μg/kg G-Pump | 1.2 μg/kg G-Pump | 2.0 μg/kg G-Pump | 0.3 μg/kg GlucaGen | 1.2 μg/kg GlucaGen | 2.0 μg/kg GlucaGen
Number analyzed (Participants) | 19 | 19 | 19 | 18 | 18 | 18
mm | 7.8 (18.9) | 18.9 (21.1) | 22.7 (25.5) | 2.2 (9.2) | 0.3 (1.0) | 0.3 (0.7)
Statistical Analysis 1: Comparison: 0.3 μg/kg G-Pump vs 0.3 μg/kg GlucaGen; Test type: Superiority or Other; p = 0.24, Mixed Models Analysis; Mean Difference (Final Values) = -6.4, 95% CI 2-sided [-17.1 to 4.3], Standard Error of Mean 5.4
Statistical Analysis 2: Comparison: 1.2 μg/kg G-Pump vs 1.2 μg/kg GlucaGen; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis; Mean Difference (Final Values) = -19.4, 95% CI 2-sided [-30.1 to -8.7], Standard Error of Mean 5.4
Statistical Analysis 3: Comparison: 2.0 μg/kg G-Pump vs 2.0 μg/kg GlucaGen; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = -23.3, 95% CI 2-sided [-34.0 to -12.6], Standard Error of Mean 5.4

10. Secondary Outcome: Infusion Site Discomfort Score at 30 Minutes
Description: Infusion site discomfort was assessed by the subject using a 100 mm Visual Analog Scale (VAS) questionnaire at 30 minutes following the initiation of dosing. Subjects were asked to draw a vertical line across the horizontal scale to indicate their current level of discomfort from 0 = no discomfort to 100 = worst possible discomfort. The distance in mm from the left hand anchor to the the first point where the subject's mark crossed the horizontal scale was measured and reported as the infusion site discomfort score.
Time Frame: At 30 minutes post-dosing
Population: All treated subjects
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0.3 μg/kg G-Pump | 1.2 μg/kg G-Pump | 2.0 μg/kg G-Pump | 0.3 μg/kg GlucaGen | 1.2 μg/kg GlucaGen | 2.0 μg/kg GlucaGen
Number analyzed (Participants) | 19 | 19 | 19 | 18 | 18 | 18
mm | 1.9 (4.8) | 1.5 (4.0) | 3.8 (9.0) | 0 (0) | 0.7 (2.6) | 0.3 (1.4)
Statistical Analysis 1: Comparison: 0.3 μg/kg G-Pump vs 0.3 μg/kg GlucaGen; Test type: Superiority or Other; p = 0.22, Mixed Models Analysis; Mean Difference (Net) = -2.0, 95% CI 2-sided [-5.1 to 1.2], Standard Error of Mean 1.6
Statistical Analysis 2: Comparison: 1.2 μg/kg G-Pump vs 1.2 μg/kg GlucaGen; Test type: Superiority or Other; p = 0.58, Mixed Models Analysis; Mean Difference (Net) = -0.9, 95% CI 2-sided [-4.0 to 2.3], Standard Error of Mean 1.6
Statistical Analysis 3: Comparison: 2.0 μg/kg G-Pump vs 2.0 μg/kg GlucaGen; Test type: Superiority or Other; p = 0.03, Mixed Models Analysis; Mean Difference (Net) = -3.6, 95% CI 2-sided [-6.7 to -0.4], Standard Error of Mean 1.6

ADVERSE EVENTS:
Time Frame: Adverse event information was collected from the time a subject provided written informed consent at the screening visit through the follow-up visit occurring 3-14 days after the final dose of study drug, a total time of 6-10 weeks per subject.
Groups:
- G-Pump™ (Glucagon Infusion): G-Pump™ (glucagon infusion); single subcutaneous doses of 0.3 μg/kg, 1.2 μg/kg and 2.0 μg/kg delivered via infusion pump
- Novo Nordisk GlucaGen®: Novo Nordisk GlucaGen®; single subcutaneous doses of 0.3 μg/kg, 1.2 μg/kg, and 2.0 μg/kg delivered by infusion pump
Arm/Group | G-Pump™ (Glucagon Infusion) | Novo Nordisk GlucaGen®
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 16/19 | 12/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | G-Pump™ (Glucagon Infusion) (N=19) | Novo Nordisk GlucaGen® (N=18)
Infusion site erythema (General disorders) | 9 (14) | 2 (2)
Infusion site swelling (General disorders) | 6 (8) | 1 (1)
Drug withdrawal headache (General disorders) | 0 (0) | 2 (2)
Infusion site bruising (General disorders) | 0 (0) | 1 (1)
Infusion site pain (General disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (6) | 6 (6)
Vomiting (Gastrointestinal disorders) | 2 (4) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Catheter site rash (General disorders) | 0 (0) | 1 (1)
Procedural dizziness (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No